CLINICAL TRIAL: NCT05270980
Title: COVID-19 Serologic Strategies for Skilled Nursing Facilities (CERO)
Brief Title: COVID-19 Serologic Strategies for Skilled Nursing Facilities
Acronym: CERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Brown University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-01281; 3U54AG063546-02S4 (NIH)
Record Dates: First submitted 2022-03-07; First posted 2022-03-08 (Actual); Results first posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Cohort Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Cohorting) (Experimental)
  Interventions: Other: Cohorting
- Control Group (No Cohorting) (No Intervention)

INTERVENTIONS:
Other: Cohorting — The cohorting strategy will result in "pairing" serology-positive staff with serology-negative residents and serology-negative staff and serology-positive residents to the degree that penetration of serologic presumed immunity allows this pairing to be positive. Any resident who refuses serology testing will be treated as if they are serology negative as the safest strategy for risk of unwanted exposure.
  Arms: Intervention Group (Cohorting)

SUMMARY:
The COVID-19 pandemic ravaged United States skilled-nursing facilities (SNFs). Novel strategies that maximize the safety and quality of life for SNF residents with ADRD and staff who care for them are urgently needed. Thus, the study's objectives are:

1. To rapidly plan and pilot test an intervention that leverages COVID-19 antibody and PCR status to pair SNF staff with residents in the safest way possible
2. To reduce reduced COVID-19 incidence rate compared to SNFs not using this novel staff-resident assignment strategy.

ELIGIBILITY:
Inclusion Criteria for Staff Stakeholders:

* Must be employees of ArchCare
* Must be members of included unit staff or those that float on those designated units
* Willing to participate in focus groups or semi-structured interviews with study team

Inclusion Criteria for Family Participants:

* Family members of residents who reside at either TCC or MMW (ArchCare facilities)
* Family member of resident who is on designated study unit or eligible to be transferred to such unit
* Willing to participate in focus groups or semi-structured interviews with study team

Inclusion Criteria for Resident Participants:

* Resident has ability to communicate and follow simple commands
* Resident has ability to communicate and follow simple commands
* English- or Spanish-speaking
* Resident has capacity to consent assessed with standard questions used to assess capacity or having a surrogate who can provide consent.
* Must agree to have serologic testing for COVID-19
* Agrees to remain on one of the facility units of study or to be transferred to such unit

Exclusion Criteria for Staff Stakeholders:

* Not employees of ArchCare
* Not members of included unit staff or those that float on those designated units
* Not willing to participate in focus groups or semi-structured interviews with study team

Exclusion Criteria for Family Participants:

* Not family members of residents who reside at either TCC or MMW (ArchCare facilities)
* Not family member of resident who is on designated study unit or eligible to be transferred to such unit
* Not willing to participate in focus groups or semi-structured interviews with study team

Exclusion Criteria for Resident Participants:

* Resident is not living in the unit of intervention
* Resident does not have ability to communicate and follow simple commands
* Not English- or Spanish-speaking
* Resident lacks capacity to consent assessed with standard questions used to assess capacity and does not have a surrogate who can provide consent.
* If resident lacks capacity, that resident does not assent with surrogate who provides assent
* Does not agree to have serologic testing for COVID-19
* Refuses to agree to remain on one of the facility units of study or to be transferred to such unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - ArchCare at Mary Manning Walsh Home (MMW), New York, New York
  - ArchCare at Terence Cardinal Cooke Health Care Center (TCC), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Joshua.Chodosh@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group (Cohorting) - Residents: Cohorting: The cohorting strategy will result in "pairing" serology-positive staff with serology-negative residents and serology-negative staff and serology-positive residents to the degree that penetration of serologic presumed immunity allows this pairing to be positive. This arm comprises residents of SNFs assigned to a cohorting strategy.
- Control Group (No Cohorting) - Residents: Residents at SNFs where no cohorting has been assigned.
- Intervention Group (Cohorting) - Staff: Staff at SNFs where the cohorting strategy has been assigned.
- Control Group (No Cohorting) - Staff: Staff at control SNFs where no cohorting strategy has been assigned.
Period: Overall Study
Arm/Group | Intervention Group (Cohorting) - Residents | Control Group (No Cohorting) - Residents | Intervention Group (Cohorting) - Staff | Control Group (No Cohorting) - Staff
Started | 14 | 2 | 50 | 21
Completed | 14 | 2 | 50 | 21
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The "Intervention Group (Cohorting) - Residents" and "Control Group (No Cohorting) - Residents" arms comprise residents at SNFs. The "Intervention Group (Cohorting) - Staff" and "Control Group (No Cohorting) - Staff" comprise staff at corresponding SNFs.
Groups:
- Control Group (No Cohorting) - Residents: Residents at SNFs where no cohorting strategy has been assigned.
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Cohorting) - Residents | Control Group (No Cohorting) - Residents | Intervention Group (Cohorting) - Staff | Control Group (No Cohorting) - Staff | Total
Number analyzed (Participants) | 14 | 2 | 50 | 21 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (13) | 61 (30) | 55 (10) | 52 (8) | 60.25 (15.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 43 | 19 | 70
  Male | 7 | 1 | 7 | 2 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 4 | 0 | 7
  Not Hispanic or Latino | 11 | 2 | 46 | 21 | 80
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 0 | 44 | 17 | 66
  White | 6 | 1 | 0 | 0 | 7
  More than one race | 3 | 0 | 5 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 2 | 50 | 21 | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of New COVID-19 Detected Infections Among Residents
Time Frame: Up to Month 5
Population: A HIPAA waiver was granted to obtain vaccination and PCR data from all residents in study units, not all of whom were participants. The overall number of participants analyzed for this outcome measure represent all residents of the SNFs for whom vaccination and PCR data were available. Therefore, the number of participants analyzed differs from the number of participants who completed the trial. Data were available for 207 residents in Intervention units and 207 residents in Control units.
Measure: Number; unit: Infections
Groups:
- Control Group (No Cohorting) - Residents: Residents of SNFs where no cohorting strategy was assigned.
Arm/Group | Intervention Group (Cohorting) - Residents | Control Group (No Cohorting) - Residents
Number analyzed (Participants) | 207 | 207
Infections | 0 | 0

2. Secondary Outcome: Number of New COVID-19 Detected Infections Among Staff
Time Frame: Up to Month 5
Population: A HIPAA waiver was granted to obtain vaccination and PCR data for all staff in study units, not all of whom were participants. The overall number of participants analyzed for this outcome measure represent all staff of the SNFs for whom vaccination and PCR data were available. Therefore, the number of participants analyzed differs from the number of participants who completed the trial. Data were available for 89 staff in Intervention units and 88 staff in Control units.
Measure: Number; unit: Infections
Arm/Group | Intervention Group (Cohorting) - Staff | Control Group (No Cohorting) - Staff
Number analyzed (Participants) | 89 | 88
Infections | 22 | 12

3. Secondary Outcome: Number of Hospitalizations Over Time
Time Frame: Up to Month 5
Population: A HIPAA waiver was granted to obtain vaccination and PCR data for all residents in study units, not all of whom were participants. The overall number of participants analyzed for this outcome measure represent all residents of the SNFs for whom vaccination and PCR data were available. Therefore, the number of participants analyzed differs from the number of participants who completed the trial. Data were available for 207 residents in Intervention units and 207 residents in Control units.
Measure: Number; unit: Hospitalizations
Groups:
- Intervention Group (Cohorting) - Residents: The cohorting strategy will result in "pairing" serology-positive staff with serology-negative residents and serology-negative staff and serology-positive residents to the degree that penetration of serologic presumed immunity allows this pairing to be positive. This arm includes residents at SNFs where cohorting has been assigned.
Arm/Group | Intervention Group (Cohorting) - Residents | Control Group (No Cohorting) - Residents
Number analyzed (Participants) | 207 | 207
Hospitalizations | 0 | 0

ADVERSE EVENTS:
Description: Deaths, serious adverse events, and non-serious adverse events were not assessed in this study.
Groups:
- Intervention Group (Cohorting) - Residents: Cohorting: The cohorting strategy will result in "pairing" serology-positive staff with serology-negative residents and serology-negative staff and serology-positive residents to the degree that penetration of serologic presumed immunity allows this pairing to be positive. Any resident who refuses serology testing will be treated as if they are serology negative as the safest strategy for risk of unwanted exposure.
Arm/Group | Intervention Group (Cohorting) - Residents | Control Group (No Cohorting) - Residents | Intervention Group (Cohorting) - Staff | Control Group (No Cohorting) - Staff
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT05270980/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT05270980/ICF_002.pdf